CLINICAL TRIAL: NCT05373797
Title: Determination of the Effect of Virtual Reality Glasses Used During Burn Dressing in Children on Parents' Satisfaction Level and Anxiety
Brief Title: The Effect of Virtual Reality Glasses Used During Burn Dressing in Children on Parents' Satisfaction Level and Anxiety
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, ümmühan kılıç, Principal Investigator, Ondokuz Mayıs University
Other Study IDs: nineteen may university; health (Other: samsun provincial health directorate)
Record Dates: First submitted 2022-04-27; First posted 2022-05-13 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-05

CONDITIONS: Randomized
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental and control group: experimental: 26 control group:26
  Interventions: Behavioral: Procedures performed on the experimental and control groups

INTERVENTIONS:
Behavioral: Procedures performed on the experimental and control groups — Intervention Group:26 Control Group (n=26):
  Other Names: experimental and control group

SUMMARY:
The study was planned as a prospective randomized controlled study and was carried out in the Training and Research Hospital burn unit outpatient clinic between 05.7.2021-1.04.2022. The population of the study consisted of the parents of children aged 5-10 years who applied to the burn unit polyclinic for dressing between the dates of the study. A total of 52 people were included in the research group. Data were collected by using the "Survey Form" consisting of 10 questions, "Newcastle Nursing Satisfaction Scale" and "Beck Anxiety Scale".

DETAILED DESCRIPTION:
In this study, the "Beck Anxiety Inventory" was applied to the parents before and after the burn dressing, while the "Newcastle Satisfaction with Nursing Scale" was applied only after dressing.

Control Group (n=26): "Parent Information Form" and "Beck Anxiety Inventory" were completed by the researcher nurse after obtaining the consent of the family and the children in the control group. After filling out the form, the parent and child were taken to the dressing room, and the researcher nurse was with both the child and the parent throughout the dressing and answered all the questions that the parent and child had. After the dressing, the child was taken to the waiting room and it was waited for the child to calm down, and "Beck Anxiety Inventory" and "Newcastle Satisfaction with Nursing Scale" were applied to the parent by the researcher nurse.

The Intervention Group (n=26): "Parent Information Form" and "Beck Anxiety Inventory" were completed by the researcher nurse after obtaining the consent of the family and the children in the intervention group. Then, the parent and child were taken to the dressing room and the child was put on virtual reality headsets and he/she watched a cartoon he/she liked. During this time, all the questions that both the child and the parent had have been answered. After the dressing, the virtual reality headsets were removed, the child was taken to the waiting room and the "Beck Anxiety Inventory" and "Newcastle Satisfaction with Nursing Scale" were applied to the parents. During all these processes, procedures were carried out in accordance with the protocols and principles established within the scope of the "COVID-19 Pandemic Measures" published by the Ministry of Health.

ELIGIBILITY:
Inclusion Criteria:

* parents
* read and write,
* understand Turkish,

Exclusion Criteria:

* under the age of 18
* do not want to participate in the study
* cannot be pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In order to determine the number of samples, power analysis was performed using the G*power program. The effect size coefficient was calculated by using the Newcastle satisfaction scale averages in source 1 (thesis), and the effect size = 0.76, and it was decided to recruit at least 26 people in each group in order to obtain 80% power at the ɑ=0.05 level, a total of 52 people in the two groups.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
The Effect of Virtual Reality Glasses Used During Burn Dressing in Children on Parents' Satisfaction Level and Anxiety | May 2022- October2022
  Using virtual reality glasses lowers parental anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Esra TURAL, PhD, Principal Investigator — omu
Locations (2):
- Turkey (Türkiye) (2):
  - Samsun Health Directorate, Samsun, İlkadım
  - 19May University, Samsun